CLINICAL TRIAL: NCT03312166
Title: First Study Evaluating Efficiency and Safety of a Compressive Device to Prevent Keloid Scars Recurrence After Surgery
Brief Title: Compressive Device to Prevent Keloïd Scars Recurrence [SCARWARS]
Acronym: SCARWARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: API/2016/75
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Keloid
Keywords: ear lobe; compression; medical device; recurrence
MeSH Terms: conditions — Keloid; Recurrence | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compression device (Experimental)
  Interventions: Device: Compression device

INTERVENTIONS:
Device: Compression device — interventions on patient are :
  * surgical excision of ear lobe keloid
  * application of compression device on sutured skin

SUMMARY:
SCARWARS study deals with the first on-human evaluation of a compressive device dedicated to the prevention of keloïd scars recurrence after surgery. The tested device is made with clinical grade silicon. SCARWARS is a monocentric study. 27 patients will be include and follow during one year. The primary outcome of this study is the number of keloid recurrence after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 yo;
* Patient with aer lobe keloid;
* Patient with an indication of reconstructive surgery;
* Signature of informed consent from the patient;
* Indication that the subject has understood the purpose and procedures required by the study and agrees to participate in the study and comply with the requirements and limitations inherent in this study;
* Patient with French social insurance.

Exclusion Criteria:

* Patient with cutaneous dermatosis or other skin pathology able to interfere with evaluated parameter (recurrence and healing quality);
* Patient with know nickel allergy;
* Patient with know silicon allergy;
* Pregnant women;
* Legal incapacity or limited legal capacity;
* Patient unlikely to cooperate in the study and / or low cooperation anticipated by the investigator;
* Patient without health insurance;
* The patient is in the period of exclusion of another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Recurrence of keloid scar | 12 month
  Recurrence will be assessed during each visit by surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Brice Chatelain, MD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No